CLINICAL TRIAL: NCT00785408
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose-ranging Study to Examine the Safety, Tolerability, and Effect on Body Weight of Subcutaneous AC2307 in Obese or Overweight Subjects
Brief Title: Study to Examine Safety, Tolerability and Effect on Body Weight of Subcutaneous AC2307 in Obese or Overweight Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFA104
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2014-12

CONDITIONS: Obesity; Overweight
Keywords: obesity; overweight; weight loss; Amylin; AC2307
MeSH Terms: conditions — Obesity; Overweight; Weight Loss | interventions — davalintide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental)
  Interventions: Drug: AC2307
- 2 (Experimental)
  Interventions: Drug: AC2307
- 3 (Experimental)
  Interventions: Drug: AC2307
- 4 (Placebo Comparator)
  Interventions: Drug: placebo
- 5 (Placebo Comparator)
  Interventions: Drug: placebo
- 6 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: AC2307 — subcutaneous, twice daily, low dose
  Arms: 1
Drug: placebo — subcutaneous, twice daily, low dose
  Arms: 4
Drug: AC2307 — subcutaneous, twice daily, middle dose
  Arms: 2
Drug: placebo — subcutaneous, twice daily, middle dose
  Arms: 5
Drug: AC2307 — subcutaneous, twice daily, high dose
  Arms: 3
Drug: placebo — subcutaneous, twice daily, high dose
  Arms: 6

SUMMARY:
A randomized, double-blind, placebo-controlled, parallel-group, dose-ranging study to examine the safety, tolerability, and effect on body weight of subcutaneous AC2307 in obese or overweight subjects.

ELIGIBILITY:
Inclusion Criteria:

- Is obese with a body mass index (BMI) ≥30 kg/m^2 to ≤45 kg/m^2, or is overweight with a BMI ≥27 kg/m^2 to <30 kg/m^2 and has at least one weight-related comorbidity (dyslipidemia, impaired fasting glucose, hypertension, obstructive sleep apnea syndrome, polycystic ovary syndrome, and/or osteoarthritis)

Exclusion Criteria:

* Has had a major change in daily physical activity (e.g., initiation of an exercise program) or has been enrolled in a weight loss program within 2 months prior to study start
* Has received AC2307 or pramlintide in a clinical study or has received prior treatment with pramlintide (SYMLIN®) or calcitonin
* Has received any investigational drug within 1 month or within a period corresponding to five times the half-life of the investigational drug, whichever is greater, before study start
* Has donated blood within 2 months before study start or is planning to donate blood during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2008-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To examine the effect on body weight of AC2307 injected subcutaneously (SC) twice daily (BID) in obese or overweight subjects | 24 weeks
To assess the safety and tolerability of AC2307 injected SC BID in obese or overweight subjects | 24 weeks

SECONDARY OUTCOMES:
To examine the effect of AC2307 injected SC BID in obese or overweight subjects on the following parameters: waist circumference; gastric emptying rate; fasting circulating metabolic parameters; patient reported outcomes | 24 weeks
To examine the pharmacokinetics of AC2307 injected SC BID in obese or overweight subjects | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Chen, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (18):
- United States (18):
  - Research Site, Birmingham, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Santa Rosa, California
  - Research Site, Walnut Creek, California
  - Research Site, Denver, Colorado
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Overland Park, Kansas
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Butte, Montana
  - Research Site, Cincinnati, Ohio
  - Research Site, Eugene, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Greer, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Olympia, Washington